CLINICAL TRIAL: NCT04112381
Title: A Pivotal Clinical Trial to Evaluate the Safety and Efficacy of Staged Bilateral Exablate Treatment of Medication Refractory Essential Tremor
Brief Title: Bilateral Treatment of Medication Refractory Essential Tremor
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET005
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Exablate Secondary Procedure (Experimental): Thalamotomy
  Interventions: Device: Exablate Model 4000 Type 1.0/1.1

INTERVENTIONS:
Device: Exablate Model 4000 Type 1.0/1.1 — Exablate thalamotomy of non tremor dominant side of the brain

SUMMARY:
The purpose of this study is to see if the MR-guided focused ultrasound (MRgFUS) thalamotomy procedure can be performed on both sides of the brain safely and effectively to reduce bilateral tremor.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 22 years or older
2. Diagnosis of medication-refractory Essential Tremor
3. Has previously underwent an Exablate index procedure in a clinical trial or in a commercial setting at least 9 months prior to enrolling in this trial
4. Able to communicate sensations during the Exablate thalamotomy procedure

Exclusion Criteria:

1. Has experienced any non-transient neurological event or worsening following the Exablate index procedure
2. Presence of unknown or MR unsafe devices anywhere in the body
3. Non-transient hemiparesis as determined by physical examination
4. Clinically significant abnormal speech function as determined by a speech pathologist
5. Pregnant or breastfeeding
6. Unstable cardiac status
7. Behavior(s) consistent with ethanol or substance abuse
8. History of bleeding disorder
9. Has received anticoagulants within one month of Exablate procedure
10. Cerebrovascular disease
11. Intracranial tumor
12. Active or suspected acute or chronic uncontrolled infection
13. Has previously had deep brain stimulation or a prior stereotactic ablation of the basal ganglia or thalamus
14. Implanted objects in the skull or the brain
15. Currently in a clinical trial involving an investigational product or non-approved use of a drug or device or in any other type of medical research
16. Unable to communicate with the investigator and staff

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Device and procedure related adverse events | 3 months
  rate of adverse events following the Exablate secondary procedure

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Stanford University, School of Medicine, Stanford, California
  - University of Maryland, Baltimore, Maryland
  - Weill Cornell Medicine, New York, New York
  - The Ohio State University - Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaplitt MG, Krishna V, Eisenberg HM, Elias WJ, Ghanouni P, Baltuch GH, Rezai A, Halpern CH, Dalm B, Fishman PS, Buch VP, Moosa S, Sarva H, Murray AM. Safety and Efficacy of Staged, Bilateral Focused Ultrasound Thalamotomy in Essential Tremor: An Open-Label Clinical Trial. JAMA Neurol. 2024 Sep 1;81(9):939-946. doi: 10.1001/jamaneurol.2024.2295. PMID 39073822